CLINICAL TRIAL: NCT05030636
Title: FIT3 : Exercise Timing for a Novel Treatment for Obesity
Brief Title: Novel Role of Exercise Timing in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie-Ève Mathieu, Marie-Ève Mathieu, Principal investigator, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERC-20-049-P
Record Dates: First submitted 2021-03-20; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Obesity, Adolescent; Exercise Timing in Obesity
Keywords: Teenagers; Exercise; Nutrition; Appetite
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Testing for each participant will comprise of 5 visits (1 preliminary and 4 experimental) conducted over a 5-8 week period at the LAPS-UdeM laboratory [Laboratoire activité physique et santé (LAPS), Université de Montréal (UdeM), Montreal, Canada]. Each participant will be assigned to the 3 different conditions in a random order. Each session will begin with 1 standard validated meal (breakfast) at 8:00 am, followed by 1 EX session (warm-up + 30 min @ 70% VO2 max + cool-down), performed at 9:30 am or 11:00 am, or no EX (30 min sedentary; Control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EX starts at 9:30 am (Experimental): A warm-up, 30 min at 70% VO2 max and a cool-down performed at 9:30 am.
  Interventions: Procedure: Acute moderate to vigorous exercise performed at a specific moment of the day
- EX starts at 11:00 am (Experimental): A warm-up, 30 min at 70% VO2 max and a cool-down performed at 11:00 am.
  Interventions: Procedure: Acute moderate to vigorous exercise performed at a specific moment of the day
- No EX (No Intervention): Control condition. A choice of 30 minutes sedentary activities.

INTERVENTIONS:
Procedure: Acute moderate to vigorous exercise performed at a specific moment of the day — Treadmill (30 minutes) at 70% of maximal aerobic capacity
  Arms: EX starts at 11:00 am; EX starts at 9:30 am

SUMMARY:
The main objective of this research project is to assess the impact of the timing of exercise on sensory perception, more specifically on taste and smell. Also, the investigators want to identify the optimal exercise timing scenario that maximizes the short-term anorexigenic effect of exercise (i.e. decrease in energy intake at the meal following the exercise session) in each group of teenagers. Hypothesis: exercise immediately before a meal (EX->MEAL) will be the most efficient scenario, and will show a larger impact on males individuals and people who suffer obesity. Subsequently, the investigators want to understand the impacts of exercise on lifestyle habits (i.e. sleep and sedentariness).

For the realization of this research project, the investigators plan to recruit approximately 144 participants, boys and girls with normal weight/obesity, aged 12 to 17 years. Of these participants, half will be male. There are two different exercise timings (i.e. performed at 9:30 am and 11:00 am using a treadmill to test the maximal aerobic capacity) and one sedentary control condition. Participants will take part in 3 experimental visits in a random order (~5 hours/visit at LAPS-UdeM + 24h of real-life monitoring). Appetite sensations, energy intake (i.e. total and macronutrient), activity monitoring using actigraphy, hormonal (i.e. anorexigenic and orexigenic) and chemosensory (i.e. cortical response to taste and smell stimulations) response will be monitored in the laboratory and/or remotely.

This project will measure acute response in laboratory and real-life settings.

DETAILED DESCRIPTION:
Obesity before adulthood is associated with increased risk of cardiometabolic disease as well as musculoskeletal and psychosocial complications. Until recently, the two major components of energy balance (i.e. energy expenditure and intake) were thought to act independently on body weight, but a growing body of knowledge in the field of human physiology supports the theory that exercise and nutrition interact (EXiNU). Complementary lifestyle behaviours [e.g. sedentariness and sleep] can also influence energy balance, all acting synergistically on energy balance (EXiNU+). Dr. Mathieu's innovative work recently revealed that the modulation of EX Timing relative to lunch can significantly improve the choice of healthier foods and lower total (-10%) and lipid (-25%) energy intake without further nutritional compensation during the rest of the day.

This unique research project focuses specifically on understanding how EX Timing can regulate energy balance, filling a major gap in the current literature. The strengths and novelty of the current proposal are that: 1) Youth of both sexes and of different body weight status will be investigated; 2) A varied profile of orexigenic and anorexigenic hormones as well as the cortical response to taste and smell will be studied to better understand food choices; 3) Sleep and sedentary behaviours will be evaluated with EX and nutrition to better assess the global influence of EX Timing on energy balance; 4) Cardiometabolic indicators linked to obesity will be monitored.

Primary objective : To identify the optimal EX Timing that maximizes the short-term anorexigenic effect of EX (i.e. decrease in energy intake at the meal following the EX session) in each group of teenagers.

Hypothesis: EX immediately before a meal (EX-->MEAL) will be the most efficient scenario, and will show a larger impact on individuals with obesity and in males.

Secondary objective #1 : To identify the optimal EX Timing that maximizes the medium-term anorexigenic effect of EX (i.e. caloric reduction during the 24 hours following the lunch) in each group of teenagers.

Hypothesis: EX immediately before a meal (EX-->MEAL) will be less efficient with time. A reduced impact on Day 1 (i.e. reduction in energy intake less important between EX and control conditions) and the absence of impact on Day 2 (similar energy intake between 4 conditions) are expected.

Secondary objective #2 : To elucidate the hormonal and chemosensory response associated with the anorexigenic effect of EX Timing.

Hypothesis: EX-->MEAL will show a maximal change in anorexigenic hormones (e.g. lowest ghrelin and highest leptin levels), and will maximally alter the cortical chemosensory processing to smell and taste. A dose-response effect is expected: the change in anorexigenic hormones being inversely proportional to the EX-meal delay.

Secondary objective #3 : Understand how complementary lifestyle factors are influenced by EX Timing and how these can induce a negative energy balance. Hypothesis: It is speculated that the EX Timing condition having the largest impact on nutrition will also reduce sedentary habits and improve sleep behaviours. Those lifestyle habits need to be monitored to control for/explore their moderating effects.

Secondary objective #4 : Monitor cardiometabolic parameters following each EX Timing scenario.

Hypothesis: The EX→Meal scenario would have larger effects on blood pressure and lipid profiles given its larger impact on energy intake. The greatest effects will be seen on participants with a poor profile (high blood pressure and lipids levels).

This project will involve 4 meetings over 4 consecutive weeks at LAPS, a laboratory equipped to meet the needs of the study [Physical Activity and Health Laboratory (FCI and don Molson) at CEPSUM].

Methods : The preliminary visit (approximately 4 hours) will include standardized questionnaires on physical activity and nutrition, various anthropometric tests (percentage of fat and body mass using DXA, height and waist circumference), an assessment of their resting metabolism (indirect calorimetry), a standardized physical test (VO2max with indirect calorimetry) as well as a culinary exposure the meals that will be served to them. During the following week (7 days), there will be a monitoring of their lifestyle (physical activity, sedentary behavior, sleep, etc.), which involves wearing an accelerometer and three food reminders by a nutritionist. Three experimental tours (approximately 5 hours / visit) will follow. These meetings present different temporal conditions in which the exercise will be immediately followed by taste and odor tests as well as blood samples. Participants will take part, in a randomized fashion, in 3 experimental conditions, all preceded by a standard breakfast served at 8 am. Condition 1: active-early (30 min at 70% VO2max) at 9 a.m., condition 2: active-late (30 min at 70% VO2max) at 11 a.m., condition 3: sedentary (control condition) from 9 a.m. to 12 p.m. Their energy intake and food choices will be assessed at 12 noon and during the 48 hours following each experimental visit, using validated lunch boxes. Measurements of appetite, taste [electroencephalogram (EEG) + gustometer] and smell (EEG + olfactometer) as well as blood tests measuring appetite hormones (ghrelin, oxytomodulin, Glucagon-Like Peptide-1 and Peptide YY-36) will be carried out at each experimental visit.

Expected outcomes : Currently, exercise periods in schools, workplaces, and free time are set randomly rather than scientifically scheduled. This is potentially suboptimal and not aligned with other medical treatments (e.g. medication) where timing is an essential component of the treatment regimen. Outcomes of this project on EX Timing will be important to improve EX interventions in order to enhance positive outcomes from each minute of exercise performed.

ELIGIBILITY:
Inclusion Criteria: Study participants :

1. must be 12-17 years old to ensure proper compliance with the study protocol and similar daily routines (i.e. attend high school);
2. have normal weight or obesity according to World Health Organisation criteria

Exclusion Criteria: Individuals will be excluded if they :

1. follow a specific diet or have food allergies;
2. have an eating disorder (e.g. anorexia or bulimia);
3. have a metabolic disease, are taking supplements or use medication that could influence the study results (e.g. insulin, lipid lowering drugs, corticosteroids);
4. are vegetarian or vegan, who cannot eat our validated meals which contain protein from animal sources;
5. have any intestinal disorders;
6. have physical limitations that restrict them from participating in our EX program;
7. are involved in competitive sports;
8. are not able to read or speak either French or English;
9. currently has COVID-19 or do not agree to respect sanitary measures during the visits; or,
10. smoke or use drugs.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Energy intake at lunch | 30 minutes
  Obtained using an ad libitum meal
Physical activity habits outside the laboratory | 24 hours
  Time spent in moderate-to-vigorous intensity.
Eating habits outside the laboratory | 24 hours
  Ambulatory monitoring of food provided that is eaten (kcal total)
Sedentary activity habits outside the laboratory | 24 hours
  Time spent in sedentary activities
Sleep activity habits outside the laboratory | 24 hours
  Time spent sleeping at night

SECONDARY OUTCOMES:
Chemosensory response - Taste | Within the 30 minutes devoted to chemosensory testing, prior to the meal at noon.
  Taste event-related potential (latency, duration and amplitude) using EEG
Circulating concentration of PYY | Within the 30 minutes devoted to chemosensory testing, prior to the meal at noon.
  orexigenic hormonal level
Chemosensory response - Smell | Within the 30 minutes devoted to chemosensory testing, prior to the meal at noon, and in the 2 hour period following meal.
  Smell event-related potential (latency, duration and amplitude) using EEG
Circulating concentration of GLP1 | Within the 30 minutes devoted to chemosensory testing, prior to the meal at noon, and in the 2 hour period following meal.
  Orexigenic hormonal level
Circulating levels of ghrelin | Within the 30 minutes devoted to chemosensory testing, prior to the meal at noon, and in the 2 hour period following meal.
  Anorexigenic hormonal levels
Oxytomodulin | Within the 30 minutes devoted to chemosensory testing, prior to the meal at noon, and in the 2 hour period following meal.
  Orexigenic hormonal levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada